CLINICAL TRIAL: NCT04360148
Title: Randomized-controlled Study for Evaluation of Ketogenic Metabolic Nutritional Pattern in Subjects With High-frequency Episodic Migraine
Brief Title: Th Effect of Ketogenic Metabolic Nutritional Pattern on High-frequency Episodic Migraine (EMIKETO)
Acronym: EMIKETO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: New Penta SRL (Industry)
Collaborators: IRCCS San Raffaele (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RP 19/23
Record Dates: First submitted 2020-04-15; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Migraine; Ketogenic Dieting; Weight Loss; Overweight; Brain Diseases
Keywords: VLCKD; migraine; diet; weight loss; ketone bodies; inflammatory state
MeSH Terms: conditions — Migraine Disorders; Weight Loss; Overweight; Brain Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Very-low-calorie-ketogenic-diet (Experimental): Very-low-calorie-ketogenic-diet (VLCKD) for 12 weeks; hypocaloric-balanced-diet (HBD)
  Interventions: Dietary Supplement: very-low-calorie-ketogenic-diet
- Hypocaloric-balanced-diet (Active Comparator): Hypocaloric-balanced-diet (HBD)
  Interventions: Other: hypocaloric-balanced-diet

INTERVENTIONS:
Dietary Supplement: very-low-calorie-ketogenic-diet — VLCKD-group will undergone to VLCKD for 8 weeks. VLCKD is based on protein preparations of high biological value. Total daily energy intake is < 800 kcal.Daily carbohydrate intake is lower than 30 g/day, while daily protein intake is approximately 1.2-1.5 g/kg of ideal body weight. The following four weeks, carbohydrates are gradually reintroduced, starting from foods with the lowest glycemic index (fruit, dairy products), followed by foods with moderate and high glycemic index (bread, pasta and cereals). The goal is to achieve a hypocaloric balanced diet (HBD), as well as the controlled group. From the 12th week to the 24 th week, all subjects enrolled will continue follow-up with HBD.
  Arms: Very-low-calorie-ketogenic-diet
Other: hypocaloric-balanced-diet — HBD-group will undergone to hypo caloric balanced diet for 24 weeks. Total daily average energy intake is 1500-1600 kcal/day. 30% of total daily energy is composed by lipids (10% MUFA, 10% PUFA, 10% SFA), 55% carbohydrates, while daily protein intake is approximately 0.8-1.5 g /kg of ideal body weight.
  Arms: Hypocaloric-balanced-diet

SUMMARY:
The study aims to investigate the impact of 2 nutritional patterns on high-frequency episodic migraine. Subjects enrolled will be randomized in two arms: a) very-low-calorie-ketogenic-diet (VLCKD), b) hypocaloric balanced non ketogenic-diet (HBD).

DETAILED DESCRIPTION:
This randomized controlled trial aims to:

* investigate the impact of very-low-calorie-ketogenic-diet (VLCKD) compared to hypocaloric balanced non ketogenic-diet (HBD) on high-frequency episodic migraine
* evaluate the impact of VLCKD or HBD on immune system, with particular regard to inflammatory and regulatory T cells
* assess aldosterone blood levels before and after VLCKD or HBD treatment The randomization will be carry out at the single center using an a proper software.

All the eligible subjects (please, see the inclusion and exclusion criteria), will be randomized in two groups. Both VLCKD or HBD will be undergone to 24 weeks of diet. For VLCKD- group, the ketogenic period will be maintained for 8 weeks. In the following four weeks, carbohydrates are gradually reintroduced, starting from foods with the lowest glycemic index (fruit, dairy products), followed by foods with moderate and high glycemic index (bread, pasta and cereals). The goal is to achieve a hypocaloric balanced diet (HBD), as well as the controlled group. From the 12th week to the 24 th week, all subjects enrolled will continue follow-up with HBD. Periodically, subjects will be monitored through physical examination (anthropometric measurements, blood pressure, heart rate, etc.) and laboratory analysis.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index >27 kg/m2
* Migraine onset <50 years with monthly frequency of 8-14 days in the last 3 months
* Absence of prophylaxis therapy for migraine in the previous 3 months
* Signing of the informed consent
* Agreement to follow all study procedures, including follow-up visits
* Negative pregnancy test, performed on urine sample
* Use of contraceptive method for all participants throughout the duration of the study
* Agreement for all study participants not to publish study information

Exclusion Criteria:

* Body mass index> 35 kg / m2;
* prophylaxis treatment for migraine in the previous 3 months
* antidepressant and neuroleptic drugs treatment during the study (including follow-up)
* non-potassium-sparing diuretics treatment during the study (including follow-up)
* Use or implantation of stimulators for migraine
* Migraine with or without excessive drug use, tension-type headache, cluster headache, sporadic or familial hemiplegic migraine, ophthalmoplegic migraine, basic migraine defined according to the ICHD-3 beta classification in the previous 3 months
* head trauma
* psychiatric diseases that can influence adherence to treatment
* Type I diabetes mellitus or type II diabetes mellitus treated with insulin therapy
* Taking supplements which affect weight
* Taking supplements containing sugars in their composition
* Pregnancy or breastfeeding
* Abuse of alcohol
* Other neurological, cardiovascular, liver, respiratory, hematologic, autoimmune diseases or alterations to laboratory tests that could compromise the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2020-02-06 (Actual); Primary Completion 2020-09-14 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in migraine frequency | at baseline (V2), at 8 weeks- the end ok ketogenic period (V5) and at 12 weeks-the end of diet (V6) and at 24 weeks -the end of follow-up (V7)
  Migraine Disability Assessment Score Questionnaire (MIDAS) is used in order to evaluate how severity migraine affects patient's life. MIDAS score: 0-25

SECONDARY OUTCOMES:
Impact of migraine episode on daily activities | at baseline (V2), at 8 weeks- the end ok ketogenic period (V5) and at 12 weeks-the end of diet (V6) and at 24 weeks -the end of follow-up (V7)
  Headache Impact Test (HIT-6) is used in order to determine how severely migraine impacts on daily activities.
  HIT-6 total score: 36-78
Weight loss | at baseline (V2), at 8 weeks- the end ok ketogenic period (V5) and at 12 weeks-the end of diet (V6) and at 24 weeks -the end of follow-up (V7)
  Physical examination will be carried out in each visit. Weight will be detected
Change in immune system parameters | at the screening (V1),at 8 weeks- the end ok ketogenic period (V5) and at 12 weeks-the end of diet (V6)
  Immune system plays a key role in overweight subjects susceptibility to inflammatory diseases. Lymphocyte subpopulation will be studied before and after VLCKD or HBD through blood tests.
Health-related quality of life | at baseline (V2), at 8 weeks- the end ok ketogenic period (V5) and at 12 weeks-the end of diet (V6)
  Health Survey-36 (SF-36) is used in order to evaluate the impact of migraine on quality of life.
  SF-36 score: The SF-36, as described in the name, is a 36-item patient-reported questionnaire that covers eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.
change in analgesic consumption | through study completion, an average of 24 weeks
  On migraine-diary, subjects will reported analgesic consumption during diet-treatment
Measure of pain | at baseline (V2), at 8 weeks- the end ok ketogenic period (V5) and at 12 weeks-the end of diet (V6)
  Visual analogue scale (VAS) is used in order to evaluate pain intensity. VAS score: 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Piero Barbanti, Prof., Principal Investigator — IRCCS San Raffaele Pisana, 00163 Rome-Italy
Locations (1):
- IRCCS San Raffaele Pisana, Rome, Italy

REFERENCES:
- [Background] GBD 2015 Neurological Disorders Collaborator Group. Global, regional, and national burden of neurological disorders during 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet Neurol. 2017 Nov;16(11):877-897. doi: 10.1016/S1474-4422(17)30299-5. Epub 2017 Sep 17. PMID 28931491
- [Background] Lipton RB, Bigal ME, Diamond M, Freitag F, Reed ML, Stewart WF; AMPP Advisory Group. Migraine prevalence, disease burden, and the need for preventive therapy. Neurology. 2007 Jan 30;68(5):343-9. doi: 10.1212/01.wnl.0000252808.97649.21. PMID 17261680
- [Background] Bigal ME, Lipton RB, Holland PR, Goadsby PJ. Obesity, migraine, and chronic migraine: possible mechanisms of interaction. Neurology. 2007 May 22;68(21):1851-61. doi: 10.1212/01.wnl.0000262045.11646.b1. PMID 17515549
- [Background] Bond DS, Roth J, Nash JM, Wing RR. Migraine and obesity: epidemiology, possible mechanisms and the potential role of weight loss treatment. Obes Rev. 2011 May;12(5):e362-71. doi: 10.1111/j.1467-789X.2010.00791.x. PMID 20673279
- [Background] Peterlin BL, Sacco S, Bernecker C, Scher AI. Adipokines and Migraine: A Systematic Review. Headache. 2016 Apr;56(4):622-44. doi: 10.1111/head.12788. Epub 2016 Mar 25. PMID 27012149
- [Background] Yumuk V, Tsigos C, Fried M, Schindler K, Busetto L, Micic D, Toplak H; Obesity Management Task Force of the European Association for the Study of Obesity. European Guidelines for Obesity Management in Adults. Obes Facts. 2015;8(6):402-24. doi: 10.1159/000442721. Epub 2015 Dec 5. PMID 26641646
- [Background] Basciani S, Costantini D, Contini S, Persichetti A, Watanabe M, Mariani S, Lubrano C, Spera G, Lenzi A, Gnessi L. Safety and efficacy of a multiphase dietetic protocol with meal replacements including a step with very low calorie diet. Endocrine. 2015 Apr;48(3):863-70. doi: 10.1007/s12020-014-0355-2. Epub 2014 Jul 26. PMID 25063307
- [Background] Ellulu MS, Patimah I, Khaza'ai H, Rahmat A, Abed Y. Obesity and inflammation: the linking mechanism and the complications. Arch Med Sci. 2017 Jun;13(4):851-863. doi: 10.5114/aoms.2016.58928. Epub 2016 Mar 31. PMID 28721154
- [Background] Lutas A, Yellen G. The ketogenic diet: metabolic influences on brain excitability and epilepsy. Trends Neurosci. 2013 Jan;36(1):32-40. doi: 10.1016/j.tins.2012.11.005. Epub 2012 Dec 8. PMID 23228828
- [Background] Klosinski LP, Yao J, Yin F, Fonteh AN, Harrington MG, Christensen TA, Trushina E, Brinton RD. White Matter Lipids as a Ketogenic Fuel Supply in Aging Female Brain: Implications for Alzheimer's Disease. EBioMedicine. 2015 Nov 3;2(12):1888-904. doi: 10.1016/j.ebiom.2015.11.002. eCollection 2015 Dec. PMID 26844268
- [Background] Paoli A, Bianco A, Damiani E, Bosco G. Ketogenic diet in neuromuscular and neurodegenerative diseases. Biomed Res Int. 2014;2014:474296. doi: 10.1155/2014/474296. Epub 2014 Jul 3. PMID 25101284
- [Background] de Almeida Rabello Oliveira M, da Rocha Ataide T, de Oliveira SL, de Melo Lucena AL, de Lira CE, Soares AA, de Almeida CB, Ximenes-da-Silva A. Effects of short-term and long-term treatment with medium- and long-chain triglycerides ketogenic diet on cortical spreading depression in young rats. Neurosci Lett. 2008 Mar 21;434(1):66-70. doi: 10.1016/j.neulet.2008.01.032. Epub 2008 Jan 19. PMID 18281154
- [Background] Bough KJ, Wetherington J, Hassel B, Pare JF, Gawryluk JW, Greene JG, Shaw R, Smith Y, Geiger JD, Dingledine RJ. Mitochondrial biogenesis in the anticonvulsant mechanism of the ketogenic diet. Ann Neurol. 2006 Aug;60(2):223-35. doi: 10.1002/ana.20899. PMID 16807920
- [Background] Mattson MP, Moehl K, Ghena N, Schmaedick M, Cheng A. Intermittent metabolic switching, neuroplasticity and brain health. Nat Rev Neurosci. 2018 Feb;19(2):63-80. doi: 10.1038/nrn.2017.156. Epub 2018 Jan 11. PMID 29321682
- [Background] Waeber C, Moskowitz MA. Migraine as an inflammatory disorder. Neurology. 2005 May 24;64(10 Suppl 2):S9-15. doi: 10.1212/wnl.64.10_suppl_2.s9. No abstract available. PMID 15911785
- [Background] Puchalska P, Crawford PA. Multi-dimensional Roles of Ketone Bodies in Fuel Metabolism, Signaling, and Therapeutics. Cell Metab. 2017 Feb 7;25(2):262-284. doi: 10.1016/j.cmet.2016.12.022. PMID 28178565
- [Background] Jeong EA, Jeon BT, Shin HJ, Kim N, Lee DH, Kim HJ, Kang SS, Cho GJ, Choi WS, Roh GS. Ketogenic diet-induced peroxisome proliferator-activated receptor-gamma activation decreases neuroinflammation in the mouse hippocampus after kainic acid-induced seizures. Exp Neurol. 2011 Dec;232(2):195-202. doi: 10.1016/j.expneurol.2011.09.001. Epub 2011 Sep 14. PMID 21939657
- [Background] Zhang Y, Xu J, Zhang K, Yang W, Li B. The Anticonvulsant Effects of Ketogenic Diet on Epileptic Seizures and Potential Mechanisms. Curr Neuropharmacol. 2018;16(1):66-70. doi: 10.2174/1570159X15666170517153509. PMID 28521671
- [Background] Kim DY, Hao J, Liu R, Turner G, Shi FD, Rho JM. Inflammation-mediated memory dysfunction and effects of a ketogenic diet in a murine model of multiple sclerosis. PLoS One. 2012;7(5):e35476. doi: 10.1371/journal.pone.0035476. Epub 2012 May 2. PMID 22567104
- [Background] Yudkoff M, Daikhin Y, Horyn O, Nissim I, Nissim I. Ketosis and brain handling of glutamate, glutamine, and GABA. Epilepsia. 2008 Nov;49 Suppl 8(Suppl 8):73-5. doi: 10.1111/j.1528-1167.2008.01841.x. PMID 19049594
- [Background] Di Lorenzo C, Curra A, Sirianni G, Coppola G, Bracaglia M, Cardillo A, De Nardis L, Pierelli F. Diet transiently improves migraine in two twin sisters: possible role of ketogenesis? Funct Neurol. 2013 Oct-Dec;28(4):305-8. PMID 24598400
- [Background] Di Lorenzo C, Coppola G, Sirianni G, Di Lorenzo G, Bracaglia M, Di Lenola D, Siracusano A, Rossi P, Pierelli F. Migraine improvement during short lasting ketogenesis: a proof-of-concept study. Eur J Neurol. 2015 Jan;22(1):170-7. doi: 10.1111/ene.12550. Epub 2014 Aug 25. PMID 25156013
- [Background] Di Lorenzo C, Coppola G, Bracaglia M, Di Lenola D, Evangelista M, Sirianni G, Rossi P, Di Lorenzo G, Serrao M, Parisi V, Pierelli F. Cortical functional correlates of responsiveness to short-lasting preventive intervention with ketogenic diet in migraine: a multimodal evoked potentials study. J Headache Pain. 2016;17:58. doi: 10.1186/s10194-016-0650-9. Epub 2016 May 31. PMID 27245682
- [Background] Fery F, Bourdoux P, Christophe J, Balasse EO. Hormonal and metabolic changes induced by an isocaloric isoproteinic ketogenic diet in healthy subjects. Diabete Metab. 1982 Dec;8(4):299-305. PMID 6761185
- [Derived] Caprio M, Moriconi E, Camajani E, Feraco A, Marzolla V, Vitiello L, Proietti S, Armani A, Gorini S, Mammi C, Egeo G, Aurilia C, Fiorentini G, Tomino C, Barbanti P. Very-low-calorie ketogenic diet vs hypocaloric balanced diet in the prevention of high-frequency episodic migraine: the EMIKETO randomized, controlled trial. J Transl Med. 2023 Oct 4;21(1):692. doi: 10.1186/s12967-023-04561-1. PMID 37794395